CLINICAL TRIAL: NCT00786110
Title: Sorafenib Plus Paclitaxel Metronomic Chemotherapy in Adreno-Cortical-Carcinoma Patients Progressing After 1st or 2nd Line Cytotoxic Chemotherapy
Brief Title: Sorafenib Plus Paclitaxel in Adreno-Cortical-Cancer Patients
Acronym: PAXO
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Turin, Italy (Other)
Responsible Party: Alfredo Berruti, Dipartimento di Scienze Cliniche e Biologiche Università di Torino
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EudraCT 2008-000759-91
Record Dates: First submitted 2008-11-05; First posted 2008-11-06 (Estimated); Last update posted 2009-02-24 (Estimated); Status verified 2009-02

CONDITIONS: Adrenocortical Carcinoma
Keywords: Sorafenib; Paclitaxel; Disease free survival
MeSH Terms: conditions — Adrenocortical Carcinoma | interventions — Sorafenib; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 arm only (Experimental): One arm only with Sorafenib plus Paclitaxel Patients enrolled will undergo strict follow-up
  Intervention: Sorafenib plus Paclitaxel
  Interventions: Drug: Sorafenib; Drug: Paclitaxel

INTERVENTIONS:
Drug: Sorafenib — Treatment scheme consisted of oral Sorafenib 400 mg p.o. bid until disease progression.
Drug: Paclitaxel — Intravenous Paclitaxel 60 mg/mq/weekly i.v., until disease progression.

SUMMARY:
The study is designed as a Phase II, prospective, non randomized, open-label, single arm, multicenter trial, in which patients with locally advanced or metastatic ACC not amenable to complete surgical resection and progressing to cytotoxic chemotherapy will receive Sorafenib plus metronomic chemotherapy as treatment.The aim of this phase II trial is to evaluate the clinical benefit and toxicity of the combination of Sorafenib plus metronomic chemotherapy in patients with locally advanced or metastatic ACC who progressed after first or second line chemotherapy.

DETAILED DESCRIPTION:
The study is designed as a Phase II, prospective, non randomized, open-label, single arm, multicenter trial, in which patients with locally advanced or metastatic ACC not amenable to complete surgical resection.

STUDY OBJECTIVES

The aim of this phase II trial is to evaluate the clinical benefit and toxicity of the combination of Sorafenib plus metronomic chemotherapy in patients with locally advanced or metastatic ACC who progressed after first or second line chemotherapy.

Primary objective

To assess the clinical benefit as measured by a non progressing rate after 4 months of the combination of Sorafenib plus weekly Paclitaxel in patients with locally advanced or metastatic ACC who progressed after first or second line chemotherapy.

Secondary objectives

* Assessment of Objective (Complete and Partial) Response Rates
* Assessment of Duration of Response
* Assessment of Hormonal Response
* Assessment of Progression-Free Survival
* Assessment of Overall Survival
* Assessment of the relationship between specific "biomarkers" and cancer- and treatment-related outcomes
* Assessment of Quality of Life by EORTC QLQ-C30
* Assessment of Toxicity

ENDPOINTS

The first disease assessment will be performed after 8-weeks, subsequent assessments will be performed every 12 weeks until end of the study.

Primary endpoint

* Progression-Free Survival rate ≥ 40% after 4 months

Secondary endpoints

* Response rate evaluation will be performed according to the RECIST criteria. The same methods of measurement and the same technique should be used to characterize each identified and reported lesion at baseline and during study.

TREATMENT SCHEME Treatment scheme consisted of oral Sorafenib 400 mg p.o. bid plus intravenous Paclitaxel 60 mg/mq/weekly i.v., until disease progression.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of ACC
* Locally advanced or metastatic disease not amenable to radical surgery resection
* Radiologically monitorable disease
* Progressing disease after one or two cytotoxic chemotherapy regimens (including a platin-based protocol)
* ECOG performance status 0-2
* Life expectancy ≥ 3 months
* Subjects with at least one uni-dimensional(for RECIST) or bi-dimensional(for WHO) measurable lesion. Lesions must be measured by CT-scan or MRI
* Age ≥ 18 years
* Adequate bone marrow reserve (neutrophils ≥ 1500/mm³ and platelets ≥ 80.000/mm³)
* Hemoglobin > 9.0 g/dl
* Total bilirubin < 1.5 times the upper limit of normal
* PT-INR/PTT < 1.5 x upper limit of normal [Patients who are being therapeutically anticoagulated with an agent such as coumadin or heparin will be allowed to participate provided that no prior evidence of underlying abnormality in these parameters exists.]
* Serum creatinine < 1.5 x upper limit of normal
* Effective contraception in pre-menopausal female and male patients
* Patient´s written informed consent
* Ability to comply with the protocol procedures

Exclusion criteria:

* History of prior malignancy, except for cured non-melanoma skin cancer, cured in situ cervical carcinoma, or other treated malignancies with no evidence of disease for at least three years.
* History of HIV infection or chronic hepatitis B or C (This criteria should be modified to allow Hepatitis B or C in protocols looking at HCC patient population)
* Active clinically serious infections (> grade 2 NCI-CTC version 3.0)
* Symptomatic metastatic brain or meningeal tumors (unless the patient is > 6 months from definitive therapy, has a negative imaging study within 4 weeks of study entry and is clinically stable with respect to the tumor at the time of study entry)
* Patients with seizure disorder requiring medication (such as steroids or anti-epileptics)
* History of organ allograft The organ allograft may be allowed as protocol specific
* Severe renal (serum creatinine > 2.5 x ULN) or hepatic insufficiency (ALT / - AST > 2.5 x ULN or ALT/AST >5 x ULN if liver function abnormalities are due to the underlying malignancy and/or total serum bilirubin > 2.5 x ULN)
* Concomitant Rifampicin
* Concomitant St. John's Wort (Hypericum perforatum)
* Warfarin is allowed; however, close monitoring of Prothrombin Time (PT) is recommended
* Decompensated heart failure (ejection fraction <45%), myocardial infarction or revascularization procedure during the last 6 months, unstable angina pectoris, uncontrolled cardiac arrhythmia
* Hypertension that cannot be controlled by medications (>160/100 mmHg despite optimal medical therapy)
* Patients with recent or active bleeding diathesis
* Pregnant or breast-feeding patients. Women of childbearing potential must have a negative pregnancy test performed within 7 days of the start of treatment.
* Both men and women enrolled in this trial must use adequate barrier birth control measures during the course of the trial and three months after the completion of trial
* Previous treatment with Sorafenib or other anticancer chemotherapy or immunotherapy during the study or within 4 weeks of study entry
* Radiotherapy during study or within 3 weeks of start of study drug. (Palliative radiotherapy will be allowed).
* Major surgery within 4 weeks of start of study
* Autologous bone marrow transplant or stem cell rescue within 4 months of study
* Use of biologic response modifiers, such as G-CSF, within 3 week of study entry. [G-CSF and other hematopoietic growth factors may be used in the management of acute toxicity such as febrile neutropenia when clinically indicated or at the discretion of the investigator, however they may not be substituted for a required dose reduction.] [Patients taking chronic erythropoietin are permitted provided no dose adjustment is undertaken within 2 months prior to the study or during the study]
* Current treatment with another investigational drug
* Any other severe acute or chronic medical or psychiatric condition, or laboratory abnormality that would impart, in the judgment of the investigator, excess risk associated with study participation or study drug administration, or which, in the judgment of the investigator, would make the patient inappropriate for entry into this study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2008-04; Primary Completion 2009-10 (Estimated); Study Completion 2010-10 (Estimated)

PRIMARY OUTCOMES:
Disease free survival | 4 months

SECONDARY OUTCOMES:
Overall survival | 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Alfredo Berruti MD, Study Chair — Internal Medicine, Department of Clinical and Biological Sciences, University of Turin, Italy; Eric Baudin, Study Director — Oncologie Endocrinienne et Médecine Nucléaire, Institut Gustave Roussy, Villejuif, France.; Massimo Terzolo, MD, Principal Investigator — Internal Medicine, Department of Clinical and Biological Sciences, University of Turin, Italy; Sophie Leboulleux, Study Director — Service de Médecine Nucléaire et de Cancérologie Endocrinienne, Institut Gustave-
Locations (5):
- Italy (5):
  - Department of Clinical and Biological Sciences, University of Turin, Orbassano
  - Azienda Ospedaliera di Padova, Padua
  - Azienda Ospedaliera Università di Palermo, Palermo
  - Policlinico Universitario Campus Biomedico- Roma, Roma
  - Ist. Clin.Humanitas, Rozzano

REFERENCES:
- [Background] Terzolo M, Angeli A, Fassnacht M, Daffara F, Tauchmanova L, Conton PA, Rossetto R, Buci L, Sperone P, Grossrubatscher E, Reimondo G, Bollito E, Papotti M, Saeger W, Hahner S, Koschker AC, Arvat E, Ambrosi B, Loli P, Lombardi G, Mannelli M, Bruzzi P, Mantero F, Allolio B, Dogliotti L, Berruti A. Adjuvant mitotane treatment for adrenocortical carcinoma. N Engl J Med. 2007 Jun 7;356(23):2372-80. doi: 10.1056/NEJMoa063360. PMID 17554118